CLINICAL TRIAL: NCT03199170
Title: Effect of Bilateral Quadratus Lumborum Block for Pain Relief in Patients With Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 817/2559(EC1)
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Caesarean Section; Spinal Anesthesia; Quadratus Lumborum Block; Analgesia
Keywords: Caesarean Section; Spinal anesthesia; Quadratus lumborum block; Postoperative pain; Intrathecal morphine
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrathecal morphine (Sham Comparator): Intrathecal morphine 0.2 mg, 0.9%NSS each side
  Interventions: Drug: Intrathecal morphine
- Intrathecal morphine with bilateral Quadratus Lumborum Block (Experimental): Intrathecal morphine 0.2 mg, 0.25%Bupivacaine 25 ml each side
  Interventions: Drug: Intrathecal morphine with bilateral Quadratus Lumborum Block
- Bilateral Quadratus Lumborum Block (Experimental): No intrathecal morphine, 0.25%Bupivacaine 25 ml each side
  Interventions: Drug: Bilateral Quadratus Lumborum Block

INTERVENTIONS:
Drug: Intrathecal morphine — 0.5% Hyperbaric bupivacaine 2 ml add morphine 0.2 mg for spinal anesthesia
  Arms: Intrathecal morphine
Drug: Bilateral Quadratus Lumborum Block — 0.25% Bupivacaine 25 ml each side for quadratus lumborum block without spinal morphine
  Arms: Bilateral Quadratus Lumborum Block
Drug: Intrathecal morphine with bilateral Quadratus Lumborum Block — 0.5% Hyperbaric bupivacaine 2 ml add morphine 0.2 mg for spinal anesthesia and 0.25% Bupivacaine 25 ml each side for quadratus lumborum block
  Arms: Intrathecal morphine with bilateral Quadratus Lumborum Block

SUMMARY:
Cesarean section commonly induces moderate to severe pain for 48 hours. These patients have additional compelling reasons to provide adequate pain relief as early mobilization is a key factor to prevent the risk of thromboembolic event which is increased during pregnancy. Beside these, patients need to be pain free to takecare for their newborn and breastfeed them. Poorly controlled pain after cesarean section also increases risk of chronic pain and postpartum depression.

Intrathecal morphine is considered the "gold standard" for postoperative pain relief after cesarean delivery. The duration of analgesic effect of morphine extend to 12-24 hours. Its widespread use is due to its favorable pharmacokinetic profile, ease of administration and low cost. Although intrathecal morphine is highly effective, its use is associated with undesirable adverse effect particularly nausea, vomiting and pruritus which reduce overall patients' satisfaction. More serious complication is the risk of delayed maternal respiratory depression.

The Quadratus Lumborum block was first described in 2007 which demonstrates a spread to the paravertebral space, thus leads to a more extensive block to T5-L1 nerve branches and a long lasting block with the potential to provide visceral pain relief. Therefore, this block has an evolving role in postoperative analgesia for many lower abdominal surgeries. As the safety is concerned, there has been one report of a patient with unilateral hip flexion and knee extension weakness leading to unplanned overnight admission following lateral quadratus lumborum block after laparoscopic gynaecological operation.

If the result favors effective, it will have the advantage of a combination with intrathecal opioid to prolong the pain free period after cesarean section which has about 4,000 cases per year.

ELIGIBILITY:
Inclusion Criteria:

* All singleton pregnant women with gestation of at least 37 weeks scheduled for elective cesarean section with American Society of Anesthesiologists (ASA) physical status 1 or 2

Exclusion Criteria:

1. refuse to receive spinal block
2. allergy to drugs used in research: morphine, local anesthetic drug and paracetamol
3. abnormal coagulopathy: congenital coagulopathy or who used anticoagulants
4. platelet dysfunction or thrombocytopenia
5. distorted anatomical structures of lumbar spines
6. systemic infection or local infection at both flank areas which are the punctures sites for quadratus lumborum block
7. unable to comprehend or use the verbal rating pain scoring system or patient-controlled analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request (PCA morphine) | 48 hours postoperatively
  Whether bilateral quadratus lumborum block can increase pain free period of patients undergo cesarean section under spinal block with intrathecal morphine or not

SECONDARY OUTCOMES:
Pain score | 48 hours postoperatively
  Pain score at rest and on movement rating by numerical rating scale in 48-hr postoperative
Requirement of rescue pain | 48 hours postoperatively
  Requirement of pain control medication
Adverse effect | 48 hours postoperatively
  Incidence of side effects e.g. nausea and vomiting, itching and sedation
Satisfaction score | 48 hours postoperatively
  Satisfaction score rated from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

REFERENCES:
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Weibel S, Neubert K, Jelting Y, Meissner W, Wockel A, Roewer N, Kranke P. Incidence and severity of chronic pain after caesarean section: A systematic review with meta-analysis. Eur J Anaesthesiol. 2016 Nov;33(11):853-865. doi: 10.1097/EJA.0000000000000535. PMID 27635953
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Triyasunant N, Chinachoti T, Duangburong S. Direct Field Block with 40 ML of 0.125% Bupivacaine in Conjunction with Intrathecal Morphine for Analgesia after Cesarean Section: A Randomized Controlled Trial. J Med Assoc Thai. 2015 Oct;98(10):1001-9. PMID 26638592
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Background] Baidya DK, Maitra S, Arora MK, Agarwal A. Quadratus lumborum block: an effective method of perioperative analgesia in children undergoing pyeloplasty. J Clin Anesth. 2015 Dec;27(8):694-6. doi: 10.1016/j.jclinane.2015.05.006. Epub 2015 Jul 11. No abstract available. PMID 26174113
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Shaaban M, Esa WA, Maheshwari K, Elsharkawy H, Soliman LM. Bilateral Continuous Quadratus Lumborum Block for Acute Postoperative Abdominal Pain as a Rescue After Opioid-Induced Respiratory Depression. A A Case Rep. 2015 Oct 1;5(7):107-11. doi: 10.1213/XAA.0000000000000188. PMID 26402020
- [Background] Wikner M. Unexpected motor weakness following quadratus lumborum block for gynaecological laparoscopy. Anaesthesia. 2017 Feb;72(2):230-232. doi: 10.1111/anae.13754. Epub 2016 Nov 28. PMID 27891579
- [Derived] Pangthipampai P, Dejarkom S, Poolsuppasit S, Luansritisakul C, Tangchittam S. Bilateral posterior Quadratus Lumborum block for pain relief after cesarean delivery: a randomized controlled trial. BMC Anesthesiol. 2021 Mar 25;21(1):90. doi: 10.1186/s12871-021-01309-6. PMID 33761894